CLINICAL TRIAL: NCT04018235
Title: An International Phase 4 Field Study to Analyse the Psychometric Properties of the Updated Module on Assessing Quality of Life of Patients With Breast Cancer (EORTC QLQ-BR23 Update- EORTCQLQ BR45)
Brief Title: Psychometric Properties of the Updated Module on Assessing Quality of Life of Patients With Breast Cancer
Acronym: EORTCQLQBR45
Status: Completed | Type: Observational
Sponsor: Helios University Hospital Wuppertal (Other)
Collaborators: Medical University of Graz (Other); Université Catholique de Louvain (Other); Hospital de Câncer de Barretos (Other); University Hospital Rijeka (Other); Evangelische Kliniken Gelsenkirchen (Unknown); University Medical Center Freiburg (Other); University Hospital Regensburg (Other); Sheba Medical Center (Other Government); Instituto Nazionale Tumori Fondazione Pascale (Unknown); Istituto Oncologico Veneto IRCCS (Other); Oslo University Hospital (Other); Jagiellonian University (Other); Oncology Department Hospital of Navarre (Unknown); University of Leeds (Other); The Netherlands Cancer Institute (Other); Tumor- und Brust-zentrum ZeTuP St. Gallen (Unknown); National Taiwan University (Other); Taipei Veterans General Hospital, Taiwan (Other Government); National Center for Global Health and Medicine, Japan (Other Government); King Hussein Cancer Center (Other); Maria Sklodowska-Curie National Research Institute of Oncology (Other); Kansai Medical University (Other); Tikur Anbessa Hospital (Unknown); Tata Memorial Hospital (Other Government); Mekelle University (Other)
Responsible Party: Sponsor
Other Study IDs: EORTC QLQ BR45
Record Dates: First submitted 2019-07-10; First posted 2019-07-12 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Breast Cancer; Quality of Life
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- localized disease or locally advanced disease: Subgroups:
  A: BCT/Ablatio + /-SN Biopsie + /- Irradiation B: BCT/Ablatio + axill Diss C: Chemotherapy D: Antihormonal Therapy E: Target Therapy
- metastatic disease: Subgroups:
  A: BCT/Ablatio + /-SN Biopsie + /- Irradiation B: BCT/Ablatio + axill Diss C: Chemotherapy D: Antihormonal Therapy E: Target Therapy F: No Surgery
- follow up disease: Subgroups:
  A: BCT/Ablatio + /-SN Biopsie + /- Irradiation B: BCT/Ablatio + axill Diss C: Chemotherapy D: Antihormonal Therapy E: Target Therapy F: No Surgery

SUMMARY:
Females breast cancer is still the most frequent type of cancer in Europe with 21 per 100,000 women .The EORTC QLQ-BR23 was one of the first modules developed to be used in conjunction with the core questionnaire EORTC QLQ-C30 and was published in 1996. Since the beginning of the work on the EORTC QLQ-BR23 some 20 years ago, much knowledge has been gathered about the epidemiology of breast cancer, and major advances have been made with regard to diagnostic and therapeutic options. Therefore, the EORTC QLG decided to update the BC23. A phase 1 to 3 module development project has been completed. This resulted in a 45 item module, retaining 23 of the original items and adding 22 new items, particularly tapping into the side effects of new systemic and local therapies.

The aim of the Phase 4 study is to test the scale structure, reliability, responsiveness to change, and validity of the EORTC QLQ-BC45 in conjunction with the EORTC QLQ- C30 in patients diagnosed with breast cancer. Participants will be enrolled in three groups according to their disease stage (1. localized disease or locally advanced disease, 2. metastatic disease, 3. follow up). Various combinations of therapies are permissible, resulting in a total of 17 subgroups.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed diagnosis of breast cancer
* no previous primary or recurrent tumour
* ability to understand the language of the questionnaire
* mental fitness to complete a questionnaire
* 18 years of age or above
* written informed consent.

Exclusion Criteria:

* no histologically confirmed diagnosis of breast cancer
* previous primary or recurrent tumour
* not mentally fit to complete a questionnaire
* not able to understand the language of the questionnaire
* younger than 18
* refusal of informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study sample will be composed of a series of consecutive cancer patients who meet the study eligibility criteria in each participating centre
Sampling Method: Non-Probability Sample
Enrollment: 576 (Actual)
Dates: Start 2019-06-14 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2021-12-17 (Actual)

PRIMARY OUTCOMES:
Psychometric Properties of the EORTC QLQ-BR45 | baseline and for some patients 1-2 weeks later (test-retest) or 3 month later (responsiveness-to-change)
  Psychometric Properties of the EORTC QLQ-BR45 (scale structure, reliability, internal consistency, responsiveness to change, and validity of the EORTC QLQ-BC45 in conjunction with the EORTC QLQ- C30 in patients diagnosed with breast cancer)

CONTACTS AND LOCATIONS:
Overall Officials: Vesna Bjelic-Radisic, Principal Investigator — Helios Universitiätsklinikum Wuppertal, Universität Witten/Herdecke
Locations (1):
- Helios Universitiätsklinikum Wuppertal, Universität Witten/Herdecke, Wuppertal, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sprangers MA, Groenvold M, Arraras JI, Franklin J, te Velde A, Muller M, Franzini L, Williams A, de Haes HC, Hopwood P, Cull A, Aaronson NK. The European Organization for Research and Treatment of Cancer breast cancer-specific quality-of-life questionnaire module: first results from a three-country field study. J Clin Oncol. 1996 Oct;14(10):2756-68. doi: 10.1200/JCO.1996.14.10.2756. PMID 8874337
- [Background] Bjelic-Radisic V, Cardoso F, Cameron D, Brain E, Kuljanic K, da Costa RA, Conroy T, Inwald EC, Serpentini S, Pinto M, Weis J, Morag O, Lindviksmoen Astrup G, Tomaszweksi KA, Pogoda K, Sinai P, Sprangers M, Aaronson N, Velikova G, Greimel E, Arraras J, Bottomley A; EORTC Quality of Life Group and Breast Cancer Group. An international update of the EORTC questionnaire for assessing quality of life in breast cancer patients: EORTC QLQ-BR45. Ann Oncol. 2020 Feb;31(2):283-288. doi: 10.1016/j.annonc.2019.10.027. Epub 2019 Dec 18. PMID 31959345